CLINICAL TRIAL: NCT03937388
Title: Effect of Gap-interleaved Stimulation Paradigms in Speech Perception Performance of Experienced Cochlear Implant Recipients: a Single-centre, Randomised Controlled Single-blinded Study
Brief Title: Speech Perception Performance With Gap-interleaved Stimulation Paradigms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angelica Perez Fornos (Other)
Collaborators: University of Innsbruck / Department of Mechatronics (Unknown)
Responsible Party: Sponsor-Investigator, Angelica Perez Fornos, Head of Engineering, Senior Lecturer, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-01938
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Deafness; Hearing Loss
Keywords: cochlear implants; electrical stimulation; processing strategy; hearing quality; speech recognition; energy consumption
MeSH Terms: conditions — Deafness; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Repeated measures, randomised, controlled, single blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear implant recipients (Experimental)
  Interventions: Other: Cochlear stimulation strategy including time-fixed gaps

INTERVENTIONS:
Other: Cochlear stimulation strategy including time-fixed gaps — Investigation of the impact of time-fixed gaps (zero-stimulation periods) in the cochlear stimulation strategy on speech performance and hearing quality.

SUMMARY:
Cochlear implants (CI) are used to help patients with severe to profound hearing loss regain auditory perception by electrical stimulation of the auditory nerve. The electrical stimulation consists of trains of charge balanced, biphasic current pulses. For each patient, individual stimulation parameters (perception threshold, most comfortable level - MCL) are determined for each electrode during fitting sessions. However, an important parameter, pulse duration, cannot be individualized for each electrode. There are certain circumstances where it would be advantageous to have the possibility of introducing variable pulse durations into the fitting strategy (e.g., optimization of energy consumption, development of combined cochleo-vestibular implants). However, since in current CI systems pulses are transmitted sequentially, introducing varying pulse widths would also introduce "gaps" (zero-stimulation periods) into the stimulation profile. The influence of such auditory gaps on speech recognition and on the quality of hearing has not been explored yet, but can be investigated in current CI users. The objective of this study is to investigate the impact of time-fixed gaps (zero-stimulation periods) in the cochlear stimulation strategy on speech performance and hearing quality.

DETAILED DESCRIPTION:
Auditory gaps can be induced in standard CI users by temporarily deactivating one to three electrodes. These gaps can be configured to have different gap durations.

The different variations of auditory stimulation with gaps will be presented to study participants via a standard MED-EL audio processor (Opus 2) bearing conformity marking. The programming of the processor will be performed using standard clinical hardware and software interfaces. These include the hardware interfaces "MAX interface box" and the "Diagnostic Interface Box" (DIB II) as well as the "MAESTRO" fitting software. After programming the respective configurations to the audio test-processor, a clinical word recognition test (Fournier) and a clinical consonant recognition test will be presented to the participants in a sound-shielded chamber using a free-field loudspeaker system.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* CI recipients using MED-EL implants (C40+, Pulsar, Sonata, Concerto, or Synchrony) and standard electrode arrays (Standard, FLEXSOFT, FLEX28, or FLEX24)
* >1 year post-implantation
* Regular CI use (at least 4 hours/day)
* At least 9 active electrodes in the device
* Good knowledge of French (at least B1 level according to the Common European Framework of Reference for Languages)

Exclusion Criteria:

* Patients with electro-acoustic stimulation (EAS) systems
* Unwillingness or inability to perform investigational tests
* Known or suspected drug or alcohol abuse
* Inability to follow the procedures of the study (e.g. due to language problems, psychological disorders, dementia, etc.)
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Performance in standardized speech perception tests | Day 1
  Consonant and word recognition tests

SECONDARY OUTCOMES:
Comparison of volume levels resulting in equal loudness perception | Day 1
  Energetic efficiency of stimulation map

OTHER OUTCOMES:
Quality of hearing | Day 1
  1-10 visual-analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Perez Fornos, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No